CLINICAL TRIAL: NCT01758159
Title: The Effect of Optimized Local Food-based Complementary Feeding With or Without Iron Supplementation on Iron Status and Gut Microbiota of 1-2 Years Old Myanmar Children
Brief Title: Effect of CFR and Iron Supplementation on Iron Status and Gut Microbiota of 1-2 Years Old Myanmar Children
Acronym: CFR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SEAMEO Regional Centre for Food and Nutrition (Other)
Collaborators: National Nutrition Center, Department of Health, Ministry of Health, Myanmar (Unknown); National Health Laboratory (Department of Health,Ministry of Health, Myanmar) (Unknown)
Responsible Party: Principal Investigator, Lwin Mar Hlaing, Medical Officer, PhD Candidate (Nutrition), SEAMEO Regional Centre for Food and Nutrition
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HHlaing CFR Myanmar
Record Dates: First submitted 2012-12-18; First posted 2013-01-01 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Iron Deficiency; Iron Deficiency Anemia
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CFR group (Experimental): The children in this group will receive complementary feeding with locally available foods according to optimized complementary feeding recommendation (CFR)
  Interventions: Dietary Supplement: Iron supplementation
- Fe group (Experimental): The children in this group will receive iron supplementation 2mg/kg/day of ferric Na EDTA (in the form of syrup) daily for 24 weeks duration.
  Interventions: Other: CFR
- CFR + Fe group (Experimental): The children in this group will receive both local food-based complementary feeding according to CFR and Iron supplementation for 24 weeks duration
  Interventions: Dietary Supplement: Iron supplementation; Other: CFR
- Control group (Placebo Comparator): The children in this group will receive basic health services and placebo syrup.

INTERVENTIONS:
Dietary Supplement: Iron supplementation
  Arms: CFR + Fe group; CFR group
Other: CFR — Complementary feeding with locally available foods according to optimized complementary feeding recommendation (CFR)
  Other Names: Complementary Feeding Recommendation
  Arms: CFR + Fe group; Fe group

SUMMARY:
Complementary feeding diet in developing countries cannot meet iron requirements of infants and young children. Iron supplementation is mostly used to treat iron deficiency whereas iron fortification is cost-effective strategy to control iron deficiency in developing countries. However, a recent study showed that iron fortification imposed negative impact on gut microbiota by increasing colonization of gut pathogen over beneficial bacteria. Gut microbiota plays essential roles in nutrient absorption, vitamin synthesis; intestinal mucosal barrier function and pathogen displacement. Iron is essential for growth and virulence of most gut pathogens and so iron supplementation might have similar negative impact on gut microbiota composition. Therefore, nutrition interventions would not be justified by assessing micronutrient status alone ignoring any possible deterioration of gut microbiota. The investigators hypothesized that optimizing the nutrient intake from locally available foods according to complementary feeding recommendation (CFR) can improve the iron status of these children while maintaining healthy gut microbiota composition.

A randomized, placebo-controlled, community-based, intervention trial will be conducted in Ayeyarwady division of Myanmar where childhood undernutrition is prevalent. The aim of this study is to compare the effect of optimized CFR to iron supplementation on iron status and gut microbiota composition of 1-2years old Myanmar children. Cluster randomization will be done at the village level to randomly allocate the villages into CFR or non-CFR villages. Individual randomization will be done to randomly assign each child into iron or placebo syrup so that individual children will receive one of 4 treatment groups (CFR, Fe, CFR + Fe, and Control) for a period of 24 weeks. Based on expected between-groups difference of hemoglobin 5g/L, at 80% power, 5% level of significance, 15% drop-out rate; after taking into account the cluster effect; required sample will be 109 per group (total = 436). A sub-sample of 15 children from each group will be randomly selected for gut microbiota assessment (total = 60). Blood samples for iron status and stool samples for gut microbiota assessment will be collected at baseline and endline. Anthropometric measurements, usual intake of iron and infectious disease morbidity will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12-18 months
* Apparently healthy
* Not consuming regular iron containing supplements during the last 4 months

Exclusion Criteria:

* With severe anemia (Hemoglobin < 50g/L)
* Malaria test positive with Immuno-chromatographic test (ICT)
* Mothers/ Caregivers are not willing to join the study
* Suffer from chronic diseases which can affect their dietary intake

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 433 (Actual)
Dates: Start 2013-02; Primary Completion 2013-08 (Actual); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Change in Iron status | Baseline (at week 0) and Endline (at week 24)
  Iron status indicators including hemoglobin (Hb), serum ferritin (SF), soluble transferrin receptor (sTfR) concentration will be measured at the beginning and at the end of 24 weeks intervention.
Change in Gut microbiota composition | Baseline (at week 0), Endline (at week 24)
  Sub-samples analysis from 60 children (15 children from each group) will be done to detect the DNA-copy number of Total bacteria, Lactobacillus, Bifidobacteria and Enterobacteria in group and Enteropathogenic E.coli (EPEC), Enterotoxigenic E.coli (ETEC) and Enteroaggregative E.coli (EAEC) species by PCR analysis at the beginning and at the end of 24 weeks intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lwin Mar Hlaing, M.B.,B.S, MPH, Principal Investigator — 1. National Nutrition Center, Ministry of Health, Myanmar. 2. South East Asian Ministers of Education Organization - Regional Center for Food and Nutrition (SEAMEO-RECFON), University of Indonesia
Locations (1):
- National Nutrition Center, Ministry of Health, Myanmar, Pan Ta Naw Township and Kyaungon Township, Ayeyarwady Region, Burma

REFERENCES:
- [Background] Santika O, Fahmida U, Ferguson EL. Development of food-based complementary feeding recommendations for 9- to 11-month-old peri-urban Indonesian infants using linear programming. J Nutr. 2009 Jan;139(1):135-41. doi: 10.3945/jn.108.092270. Epub 2008 Dec 3. PMID 19056658
- [Background] Ferguson EL, Darmon N, Fahmida U, Fitriyanti S, Harper TB, Premachandra IM. Design of optimal food-based complementary feeding recommendations and identification of key "problem nutrients" using goal programming. J Nutr. 2006 Sep;136(9):2399-404. doi: 10.1093/jn/136.9.2399. PMID 16920861
- [Background] Fahmida U, Preedy VR. Food-Based Complementary Feeding and Its Impact on Growth: Southeast Asian Perspectives, Handbook of Growth and Growth Monitoring in Health and Disease. Springer New York; 2012. p. 1599-610.
- [Background] Gibson RS, Anderson VP. A review of interventions based on dietary diversification or modification strategies with the potential to enhance intakes of total and absorbable zinc. Food Nutr Bull. 2009 Mar;30(1 Suppl):S108-43. doi: 10.1177/15648265090301S107. PMID 19472604
- [Background] Gibson RS, Ferguson EL, Lehrfeld J. Complementary foods for infant feeding in developing countries: their nutrient adequacy and improvement. Eur J Clin Nutr. 1998 Oct;52(10):764-70. doi: 10.1038/sj.ejcn.1600645. PMID 9805226
- [Background] Zimmermann MB, Hurrell RF. Nutritional iron deficiency. Lancet. 2007 Aug 11;370(9586):511-20. doi: 10.1016/S0140-6736(07)61235-5. PMID 17693180
- [Background] Iannotti LL, Tielsch JM, Black MM, Black RE. Iron supplementation in early childhood: health benefits and risks. Am J Clin Nutr. 2006 Dec;84(6):1261-76. doi: 10.1093/ajcn/84.6.1261. PMID 17158406
- [Background] World Health Organization. Conclusions and recommendations of the WHO Consultation on prevention and control of iron deficiency in infants and young children in malaria-endemic areas. Food Nutr Bull. 2007 Dec;28(4 Suppl):S621-7. doi: 10.1177/15648265070284s414. No abstract available. PMID 18297899
- [Background] Prakash S, Rodes L, Coussa-Charley M, Tomaro-Duchesneau C. Gut microbiota: next frontier in understanding human health and development of biotherapeutics. Biologics. 2011;5:71-86. doi: 10.2147/BTT.S19099. Epub 2011 Jul 11. PMID 21847343
- [Background] Zimmermann MB, Chassard C, Rohner F, N'goran EK, Nindjin C, Dostal A, Utzinger J, Ghattas H, Lacroix C, Hurrell RF. The effects of iron fortification on the gut microbiota in African children: a randomized controlled trial in Cote d'Ivoire. Am J Clin Nutr. 2010 Dec;92(6):1406-15. doi: 10.3945/ajcn.110.004564. Epub 2010 Oct 20. PMID 20962160
- [Background] Monira S, Nakamura S, Gotoh K, Izutsu K, Watanabe H, Alam NH, Endtz HP, Cravioto A, Ali SI, Nakaya T, Horii T, Iida T, Alam M. Gut microbiota of healthy and malnourished children in bangladesh. Front Microbiol. 2011 Nov 21;2:228. doi: 10.3389/fmicb.2011.00228. eCollection 2011. PMID 22125551
- [Background] Yap GC, Chee KK, Hong PY, Lay C, Satria CD, Sumadiono, Soenarto Y, Haksari EL, Aw M, Shek LP, Chua KY, Zhao Y, Leow D, Lee BW. Evaluation of stool microbiota signatures in two cohorts of Asian (Singapore and Indonesia) newborns at risk of atopy. BMC Microbiol. 2011 Aug 26;11:193. doi: 10.1186/1471-2180-11-193. PMID 21875444